CLINICAL TRIAL: NCT07097454
Title: Effectiveness of Hypotension Prediction Index (HPI) in Preventing Hypotension in the Post-Anesthesia Care Unit (PACU): A Prospective, Randomized, Controlled Trial
Brief Title: Effectiveness of Hypotension Prediction Index (HPI) in Preventing Hypotension in the Post-Anesthesia Care Unit (PACU)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wonkwang University Hospital (Other)
Responsible Party: Principal Investigator, Cheol Lee,MD,PhD,, Professor, Wonkwang University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WonkwangUH21
Record Dates: First submitted 2025-07-15; First posted 2025-07-31 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Hypotension; Postoperative Complications
Keywords: Hypotension Prediction Index (HPI); PACU; Hemodynamic Monitoring; Arterial Pressure Waveform; HemoSphere
MeSH Terms: conditions — Hypotension; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Two-arm, parallel, randomized controlled trial comparing HPI-guided monitoring versus standard care in the PACU.
Masking Description: No masking; open-label study due to the nature of real-time hemodynamic monitoring intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- HPI-guided Monitoring (Experimental): Participants in this group will receive continuous Hypotension Prediction Index (HPI) monitoring using the Edwards Lifesciences HemoSphere platform. Interventions such as fluid boluses or vasopressors will be administered when HPI ≥ 85, following institutional protocols.
  Interventions: Device: Hypotension Prediction Index Monitoring
- Control Group (Active Comparator): Participants in this group will receive standard post-anesthesia care unit (PACU) monitoring, including non-invasive blood pressure, heart rate, and oxygen saturation. Interventions will follow usual care without guidance from HPI.
  Interventions: Other: Standard PACU Monitoring

INTERVENTIONS:
Device: Hypotension Prediction Index Monitoring — HPI monitoring is performed using the Edwards Lifesciences HemoSphere platform to provide real-time hypotension prediction based on arterial pressure waveform analysis. Interventions such as fluid bolus or vasopressor are administered per protocol when HPI ≥ 85.
  Other Names: HPI Monitoring
  Arms: HPI-guided Monitoring
Other: Standard PACU Monitoring — Standard monitoring in the post-anesthesia care unit (PACU), including non-invasive blood pressure, heart rate, and oxygen saturation measurements. No Hypotension Prediction Index (HPI) monitoring is used. Interventions are performed according to routine institutional practices.
  Other Names: Usual Care
  Arms: Control Group

SUMMARY:
Postoperative hypotension in the post-anesthesia care unit (PACU) is common and linked to adverse outcomes. The Hypotension Prediction Index (HPI) predicts hypotensive events intraoperatively, but its PACU application is unexplored. This study aims to investigate the effectiveness of HPI-guided monitoring in preventing PACU hypotension.

DETAILED DESCRIPTION:
Study Design This prospective, randomized, controlled, single-center trial will be conducted in the PACU of a tertiary care hospital. The study aims to evaluate the effectiveness of HPI in preventing postoperative hypotension. All procedures follow institutional protocols, and the trial is designed to reduce bias through randomization and stratification.

Study Population Eligible patients are adults (≥ 19 years) undergoing elective surgery under general anesthesia, with arterial catheters in place and an expected PACU stay of ≥ 30 minutes. Exclusion criteria include immediate postoperative ICU admission, use of vasopressors during anesthesia emergence, ASA physical status V, or contraindications to arterial monitoring. These criteria ensure a focus on patients suitable for PACU monitoring with arterial lines. The study population is representative of high-risk surgical patients requiring advanced hemodynamic monitoring.

Intervention Patients will be randomized 1:1 to the HPI group, which receives continuous HPI monitoring (Edwards Lifesciences HemoSphere platform, Irvine, CA, USA) with interventions such as fluid boluses or vasopressors if HPI is ≥ 85 per protocol, or to the control group, which receives standard PACU monitoring including non-invasive blood pressure, heart rate, and oxygen saturation. The interventions in the HPI group follow institutional guidelines to ensure consistency, while the control group receives routine PACU monitoring practices. Randomization will be used in a computer-generated sequence, stratified by ASA class (I-II vs. III-IV) to balance risk profiles.

Outcomes The primary outcome is the incidence of hypotension (mean arterial pressure [MAP] < 65 mmHg for more than 1 minute) during the PACU stay. Secondary outcomes include time to the first hypotensive episode, total duration of hypotension, vasopressor and fluid administration (frequency and dose), PACU stay duration, and postoperative complications such as nausea and acute kidney injury. Acute kidney injury (AKI) in the PACU was defined using the Kidney Disease: Improving Global Outcomes (KDIGO) criteria, specifically as an increase in serum creatinine by ≥ 0.3 mg/dL within 48 hours of surgery or an increase to ≥1.5 times baseline within 7 days, assess via blood samples collect during or immediately after the PACU stay. Urine output criteria are not used due to the short PACU duration and inconsistent catheterization. These outcomes are selected to evaluate both the effectiveness and impact of the HPI on clinical management. Complications are monitored to assess safety and secondary effects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 19 years
* Undergoing elective surgery under general anesthesia
* Presence of intra-arterial catheter at the end of surgery
* Expected PACU stay of ≥ 30 minutes
* Provided written informed consent

Exclusion Criteria:

* Immediate postoperative ICU admission
* Use of vasopressors during emergence from anesthesia
* ASA physical status classification of V
* Known contraindications to arterial line placement
* Participation in another interventional study within 30 days

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2025-05-06 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-07-11 (Actual)

PRIMARY OUTCOMES:
Incidence of Postoperative Hypotension in the PACU | From PACU admission to discharge, typically within 90 minutes
  Defined as mean arterial pressure (MAP) < 65 mmHg lasting for more than 1 minute during the patient's stay in the post-anesthesia care unit (PACU).

SECONDARY OUTCOMES:
Time to First Hypotensive Episode | From PACU admission until first hypotensive event
  Time elapsed from PACU admission to the first hypotensive episode (MAP < 65 mmHg for >1 minute).
Vasopressor Use | From PACU admission until first hypotensive episode, assessed up to 2 hours
  Percentage of patients receiving any vasopressor during PACU stay.
PACU Length of Stay | Duration of PACU stay, typically 30 to 90 minutes
  Total duration (in minutes) of PACU stay.
Incidence of Postoperative Complications | Within 24 hours after PACU admission
  Occurrence of postoperative complications during PACU stay, including nausea/vomiting and acute kidney injury as defined by KDIGO criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Cheol Lee, M.D.,Ph.D, Principal Investigator — Department of anesthesiology and pain medicine, Wonkwang University Hospital
Locations (1):
- Wonkwag UH, Iksan, Jeollabukdo, South Korea

IPD SHARING:
Plan to Share IPD: No